CLINICAL TRIAL: NCT06503406
Title: A Prospective Study Using SupraSDRM® in Promoting Healing and Reducing the Time to Grafting of Full-thickness Wounds
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Metis Foundation (Other)
Collaborators: The University of Texas Medical Branch, Galveston (Other); United States Department of Defense (U.S. Federal Agency); The United States Army Institute of Surgical Research (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00076270; CDMRP-RC220169 (Other Grant/Funding Number: Congressionally Directed Medical Research Program); E04634.1a (Other: Office of Human and Animal Research Oversight)
Record Dates: First submitted 2024-07-01; First posted 2024-07-16 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Surgical Wound; Burns; Trauma Injury
MeSH Terms: conditions — Surgical Wound; Burns; Accidental Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SupraSDRM® (Experimental): Once randomization is completed and the site is adequately debrided the assigned treatment dressing will be applied according to their respective instructions for use. Supplemental supportive dressings including negative pressure treatment may be used in conjunction with the study dressings.
  Interventions: Device: SupraSDRM®
- SOC Skin Substitute (Active Comparator): Once randomization is completed and the site is adequately debrided the assigned treatment dressing will be applied according to their respective instructions for use. Supplemental supportive dressings including negative pressure treatment may be used in conjunction with the study dressings.
  Interventions: Device: NovoSorb® BTM

INTERVENTIONS:
Device: SupraSDRM® — SupraSDRM® Bidegradable Matrix Wound Dressing is a tri-polymber, Biodegrable dermal covering manufactured by PolyMedics Innovations, GmbH.
  Arms: SupraSDRM®
Device: NovoSorb® BTM — NovoSorb® BTM absorbable synthetic wound dressing, PolyNovo Biomaterials, K172140
  Arms: SOC Skin Substitute

SUMMARY:
This is a prospective, randomized, controlled, multi-center clinical study comparing SupraSDRM® to standard of care wound dressing, BTM, in the treatment of full-thickness wounds deemed not immediately suitable for definitive grafting will be performed.

DETAILED DESCRIPTION:
Twenty-four patients with full-thickness wounds fulfilling inclusion criteria of the study will be consented and enrolled into the clinical trial. An area (≥ 5 and ≤125 cm2) deemed not immediately ready to accept skin graft will be designated as the study site. The study site will be randomized to receive either SupraSDRM® or the SoC wound dressing, NovoSorb® BTM.

ELIGIBILITY:
Inclusion Criteria:

* Patient age ≥18 years and ≤85 years
* Full-thickness traumatic injury, surgical wound, or excised full-thickness burn (e.g., friction, contact, flame, scalding etiology), where immediate grafting is not deemed suitable by the treating surgeon
* Wound size ≥ 5cm2 not immediately suitable for graft application
* Subject or legally authorized representative is able and willing to sign informed consent

Exclusion Criteria:

* Study wound may not include areas of the face, and neck and genitalia.
* Wound with metal hardware exposure
* Pressure sores
* Wounds with residual malignancy
* Wound infection at the time of planned wound dressing application
* Wound that is a part of an active treatment arm of an interventional study (within 90 days of Screening Visit)
* Pregnancy/lactation
* Subjects who are unable to follow the protocol or who are likely to be non-compliant
* Subjects with uncontrolled diabetes (defined by Hgb A1C >10)
* Subjects who are receiving systemic steroids or immune suppressive treatment
* Subject with a known allergy to polylactide, polycaprolactone, polyvinyl alcohol, trimethylene carbonate or resorbable suture materials.
* Prisoners

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Number of days between the application of the dermal substitute to when the dermal substitute is deemed suitable for grafting by the treatment care team. | up to 5 weeks
  This endpoint is based on the ability of the dermal substitute to rapidly vascularize and allow for placement of a skin graft.

SECONDARY OUTCOMES:
Clinical incidence of skin substitute infection | up to 5 weeks
  Incidence of infections and inflammatory response and scar development
Days of skin graft application from time of SupraSDRM® or SoC application | up to 5 weeks
  The wounds will be assessed for their readiness for grafting by their treating surgeon at minimum weekly
Percentage graft survival as assessed 7 days after skin graft application | 7 days
  Percent of graft survival will be measured by clinical assessment
Number of return trips to the OR | up to 1 year
  The wounds will be assessed by their care team as part of standard care procedures. Research personal will document any areas of concern or additional surgeries required.
Skin graft contraction | up to 1 year
  Patient and Observer Scar Assessment Scale (POSAS) Questionnaire will be used to assess scaring and contraction. This scale uses a 1-10 rating scale with 1 being normal and 10 being worst imaginable outcome.
Wound Pain scale 1-10 | up to 1 year
  Patients will be asked to rate their pain 0-10 (0=no pain and 10=a lot of pain) at each visit
Cost-effectiveness | up to 1 year
  looking at the overall length of stay in the hospital, the number of trips to the operating room and cost of skin substitute will help determine if the study dressing is more or less cost affective

CONTACTS AND LOCATIONS:
Overall Officials: Rodney Chan, MD, Principal Investigator — Metis Foundation

IPD SHARING:
Plan to Share IPD: No